CLINICAL TRIAL: NCT06242470
Title: A Phase 1/1b First-in-Human, Open Label, Dose Escalation and Cohort Expansion Study of MGC026 in Participants With Advanced Solid Tumors
Brief Title: A Study of MGC026 in Participants With Advanced Solid Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: MacroGenics (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CP-MGC026-01
Record Dates: First submitted 2024-01-12; First posted 2024-02-05 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Advanced Solid Tumor; Advanced Cancer; Metastatic Cancer; Squamous Cell Carcinoma of Head and Neck; Non Small Cell Lung Cancer; Small-cell Lung Cancer; Bladder Cancer; Sarcoma; Endometrial Cancer; Melanoma; Castration Resistant Prostatic Cancer; Cervical Cancer; Colorectal Cancer; Gastric Cancer; Gastro-esophageal Cancer; Pancreas Cancer; Clear Cell Renal Cell Carcinoma; Hepatocellular Carcinoma; Platinum-resistant Ovarian Cancer; Breast Cancer; Ovarian Cancer; Esophageal Squamous Cell Cancer (SCC)
MeSH Terms: conditions — Neoplasm Metastasis; Squamous Cell Carcinoma of Head and Neck; Carcinoma, Non-Small-Cell Lung; Small Cell Lung Carcinoma; Urinary Bladder Neoplasms; Sarcoma; Endometrial Neoplasms; Melanoma; Prostatic Neoplasms, Castration-Resistant; Uterine Cervical Neoplasms; Colorectal Neoplasms; Stomach Neoplasms; Pancreatic Neoplasms; Carcinoma, Renal Cell; Carcinoma, Hepatocellular; Breast Neoplasms; Ovarian Neoplasms; Esophageal Squamous Cell Carcinoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (12):
- Cohort 1 (Experimental): MGC026 is a topoisomerase 1 inhibitor (TOP1i)-based ADC that targets B7-H3 administered IV every 3 weeks.
  Interventions: Biological: MGC026 Dose Escalation
- Cohort 2 (Experimental)
  Interventions: Biological: MGC026 Dose Escalation
- Cohort 3 (Experimental)
  Interventions: Biological: MGC026 Dose Escalation
- Cohort 4 (Experimental)
  Interventions: Biological: MGC026 Dose Escalation
- Cohort 5 (Experimental)
  Interventions: Biological: MGC026 Dose Escalation
- Cohort 6 (Experimental)
  Interventions: Biological: MGC026 Dose Escalation
- Expansion cohort 1 (Experimental)
  Interventions: Biological: MGC026 Dose for Expansion
- Expansion cohort 2 (Experimental)
  Interventions: Biological: MGC026 Dose for Expansion
- Expansion cohort 3 (Experimental)
  Interventions: Biological: MGC026 Dose for Expansion
- Expansion cohort 4 (Experimental)
  Interventions: Biological: MGC026 Dose for Expansion
- Expansion Cohort 5 (Experimental)
  Interventions: Biological: MGC026 Dose for Expansion
- Expansion Cohort 6 (Experimental)
  Interventions: Biological: MGC026 Dose for Expansion

INTERVENTIONS:
Biological: MGC026 Dose Escalation — Escalating doses of MGC026
  Arms: Cohort 1; Cohort 2; Cohort 3; Cohort 4; Cohort 5; Cohort 6
Biological: MGC026 Dose for Expansion — MGC026 recommended dose for expansion
  Arms: Expansion Cohort 5; Expansion Cohort 6; Expansion cohort 1; Expansion cohort 2; Expansion cohort 3; Expansion cohort 4

SUMMARY:
The study is designed to understand the safety, tolerability, pharmacokinetics, immunogenicity, and preliminary antitumor activity of MGC026 in participants with relapsed or refractory, unresectable, locally advanced or metastatic solid tumors The study has a dose escalation portion and a cohort expansion portion of the study.

Participants will receive MGC026 by intravenous (IV) infusion. The dose of MGC026 will be assigned at the time of enrollment. Participants may receive up to 35 treatments if there are no severe side effects and as long as the cancer does not get worse. Participants will be monitored for side effects, and progression of cancer, have blood samples collected for routing laboratory work, and blood samples collected for research purposes.

ELIGIBILITY:
Inclusion Criteria:

* Adults ≥ 18 years old, able to provide informed consent
* Adequate performance and laboratory parameters
* Availability of archival or formalin-fixed paraffin-embedded tumor tissue sample. Participants may undergo a fresh tumor biopsy to obtain a specimen for testing if an archival tumor sample is not available. Participants with no available archival tissue sample who cannot safely undergo a fresh biopsy as determined by consultation between the sponsor and investigator are eligible
* Unresectable, locally advanced or metastatic solid tumors including: squamous cell cancer (SCC) of the head and neck, esophageal SCC, squamous and non-squamous non-small cell lung cancer, small cell lung cancer, bladder cancer, sarcoma, endometrial cancer, melanoma, castration resistant prostate cancer, breast cancer, ovarian cancer, cervical cancer, colorectal cancer gastric or gastroesophageal cancer, pancreatic carcinoma, clear cell renal cell cancer or hepatocellular cancer.
* Measurable disease per RECIST v1.1. Participants with metastatic CRPC without measurable disease are eligible.
* Must be willing to use highly effective methods of birth control from the time of consent through 7 months after discontinuation of MGC026.
* Not pregnant or breastfeeding.

Exclusion Criteria:

* Any underlying medical or psychiatric condition impairing participant's ability to receive, tolerate, or comply with the planned treatment or study procedures.
* Another cancer that required treatment within the past 2 years, with the exception of those with low risk of cancer spreading or death such as adequately treated non melanomatous skin cancer, localized prostate cancer (Gleason Score < 6), or carcinoma in situ.
* Patients with history of prior central nervous system (CNS) metastasis must have been treated, be asymptomatic, and not have concurrent treatment for CNS disease, progression of CNS metastases on magnetic resonance imaging, computed tomography or positron emission tomography, or history of leptomeningeal disease or cord compression at the time of enrollment.
* Treatment with surgery, systemic cancer therapy, immunotherapy, chimeric antigen receptor-T therapy, or anti-hormonal within protocol specified intervals.
* Prior treatment with any B7-H3 targeted agent for cancer or any ADC with a topoisomerase payload.
* Prior autologous or allogeneic stem cell or solid organ transplant.
* Clinically significant cardiovascular, pulmonary, or gastrointestinal disorders.
* Active viral, bacterial, or systemic fungal infection requiring parenteral treatment within 1 week of first study drug administration.
* Known history of hepatitis B or C infection or known positive test for hepatitis B surface antigen or core antigen, or hepatitis C polymerase chain reaction.
* Known positive testing for human immunodeficiency virus or history of acquired immune deficiency syndrome.
* History of primary immunodeficiency.
* Major trauma or major surgery within 4 weeks of first study drug administration.
* Known hypersensitivity to recombinant proteins.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2024-03-06 (Actual); Primary Completion 2028-05 (Estimated); Study Completion 2028-10 (Estimated)

PRIMARY OUTCOMES:
Number of participants with adverse events (AEs) and serious AEs (SAEs), AEs leading to dose delay, AEs leading to dose reduction, AEs leading to treatment discontinuations, AEs meeting criteria for dose limiting toxicity, and AEs of special interest. | Throughout the study, up to 135 weeks

SECONDARY OUTCOMES:
Overall response rate in advanced solid tumors | Throughout the study, up to 135 weeks
  The objective response rate (ORR) per Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST 1.1) is used to estimate the proportion of participants in the Response Evaluable population who achieve best overall response of complete response (CR) or partial response (PR) (called responders).
  Complete response (CR) is defined as disappearance of all target and non-target lesions.
  Partial response (PR) is defined as at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters, no progression of non-target lesions, and no new lesions
Duration of response (DoR) in advanced solid tumors | Throughout the study, up to 135 weeks
  DoR is defined as the time from the date of initial response (CR or PR) to the date of first documented progression or death from any cause, whichever occurs first. (RECIST 1.1) is used to classify responses.
ORR rate in metastatic castration resistant prostate cancer (mCRPC) | Throughout the study, up to 135 weeks
  The ORR per Prostate Cancer Working Group 3 (PCWG3) criteria is estimated as the proportion of participants in the Response Evaluable population who achieve best overall response of CR or PR (called responders).
DoR in mCRPC | Throughout the study, up to 135 weeks
  DoR is defined as the time from the date of initial response (CR or PR) to the date of first documented progression, per PCWG3 criteria or death from any cause, whichever occurs first.
Mean (standard deviation [SD]) of MGC026 total and conjugated antibody maximum serum concentration (Cmax) | Cycle 1 Day 1: at baseline, end of infusion (EOI) approximately 1 hr, 4hrs after EOI, Day 2 and Day 4.
  The maximum concentration in the bloodstream at the end of the infusion.
Mean (standard deviation [SD]) of MGC026 unconjugated payload Cmax | Cycle 1 Day 1: at baseline, end of infusion (EOI) approximately 1 hr, 4hrs after EOI, Day 2 and Day 4.
  The maximum concentration in the bloodstream at the end of the infusion.
Mean (SD) of MGC026 total and conjugated antibody area under the time concentration curve (AUC) | Cycle 1 Day 1: at baseline, EOI approximately 1 hr, 4hrs after EOI, Day 2, Day 4, Day 8, Day 15, and predose Cycle 2 Day 1
  Calculated exposure to MGC026
Mean (SD) of MGC026 unconjugated payload AUC | Cycle 1 Day 1: at baseline, EOI approximately 1 hr, 4hrs after EOI, Day 2, Day 4, Day 8, Day 15, and predose Cycle 2 Day 1
  Calculated exposure to MGC026
Number of participants who develop anti-MGC026 antibodies (immunogenicity) | Day 1, Day 15, and Day 1 of every 21-day cycle, throughout the study, average of 1 year.
  Development of anti-MGC026 antibodies in the bloodstream

CONTACTS AND LOCATIONS:
Overall Officials: Denise Casey, MD, Study Director — MacroGenics
Locations (12):
- United States (7):
  - The Angeles Clinic and Research Institute, Los Angeles, California
  - START Midwest, Grand Rapids, Michigan
  - START-New York Long Island, Lake Success, New York
  - Providence Cancer Institute, Portland, Oregon
  - The University of Texas MD Anderson Cancer Center, Houston, Texas
  - University of Texas Health Science Center at Houston, Houston, Texas
  - START Mountain Region, West Valley City, Utah
- Australia (3):
  - ICON Cancer Centre Wesley, Auchenflower, Queensland
  - ICON Cancer Centre Kurralta Park, Kurralta Park, South Australia
  - Austin Health- Olivia Newton John Cancer Center, Heidelberg, Victoria
- United Kingdom (2):
  - Oxford University Hospitals NHS Foundation Trust, Oxford
  - The Royal Marsden NHS Foundation Trust, Sutton

IPD SHARING:
Plan to Share IPD: No